CLINICAL TRIAL: NCT05014763
Title: Comparison of Peri-implant Tissue Stability Following Soft Tissue Augmentation Harvested From the Deep Palate or the Tuberosity Area: A Randomized Controlled Clinical Trial
Brief Title: Peri-implant Tissue Stability Following Tissue Augmentation Harvested From Deep Palate or Tuberosity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9811213001
Record Dates: First submitted 2021-07-26; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Alveolar Ridge Augmentation; Tissue Transplantation; Tissue Donors

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTG from deep palate (Active Comparator): The connective tissue graft harvested from the deep palate during flap elevation for implant placement
  Interventions: Procedure: connective tissue graft
- CTG from tuberosity (Experimental): The connective tissue graft harvested from the tuberosity
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Procedure: connective tissue graft — Connective tissue graft surgery will be done for increasing soft tissue volume. In this methods connective tissue will be harvested from lateral palate or tuberosity area.

SUMMARY:
This study will compare peri implant tissue stability following connective tissue graft harvested fromLateral Palate or the Tuberosity Area. As far as we know, it remains controversial whether peri-implant soft tissue stability could be achieved after soft tissue augmentation with the connective tissue graft from the tuberosity or the lateral palate. Soft tissue stability evaluated by intra oral scanner will be described as primary outcome.

DETAILED DESCRIPTION:
Ridge resorption is a common finding after tooth extraction. Recently, there is an increasing concern about this issue during implant-supported reconstruction in the esthetic zone. Although the previous studies supports the guided bone regeneration procedures for reconstruction of contour deficiencies, the replacement of the mineralized materials with the bone has been questioned. Therefore, recently, using connective tissue grafts instead of allogenic or xenogenic materials has been addressed.

The palate is routinely used as the donor site for harvesting the connective tissue graft. The graft can be harvested by de-epithelialized method or it can be harvested conventionally from deep palate during flap elevation. Another choice for harvesting the connective tissue graft is the tuberosity area, which can be used when you need small to moderate amount of soft tissue (around 1-2 implants). The connective tissues harvested from these sites have quite different characteristics, which might influence on the fate of the treatment in terms of the stability.

therefore, we decided to compare the stability of the grafts harvested from the deep palate or tuberosity.

ELIGIBILITY:
Inclusion Criteria:

1. more than 18 years old.
2. systemically and periodontally healthy patients.
3. need of single implant placement between two maxillary teeth.
4. need of tissue augmentation due to concavity or soft tissue thickness less than 2 millimetres .
5. more than 3 month after extraction.
6. full mouth plaque index lesser than 20%.
7. sufficient mesiodistal and buccolingual space.
8. At least 10 millimetres mesiodistal dimension in tuberosity.
9. sufficient implant primary stability.
10. at least 6 mm crestal ridge width.

Exclusion Criteria:

1. History of periodontitis and radiotherapy.
2. Need of horizontal ridge augmentation.
3. Previous soft tissue augmentation.
4. Heavy smoker( more than 10 cigarette per day)
5. Local or systemic conditions that would interfere with routine periodontal therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
soft tissue volume change 0-3 | from baseline (immediately before surgery) to 3 months
  changes of soft tissue volume from baseline (immediately before surgery) to 3 months by intra oral scanner
soft tissue volume change 0-6 | from baseline (immediately before surgery) to 6 months
  changes of soft tissue volume from baseline (immediately before surgery) to 6 months by intra oral scanner
soft tissue volume change 3-6 | from 3 months to 6 months
  changes of soft tissue volume from 3 months to 6 months by intra oral scanner

SECONDARY OUTCOMES:
The level of the pain by questionnaire through visual analogue scale | immediately after surgery
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 1
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 2
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 3
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 4
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 5
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 6
  evaluation of the level of the pain by questionnaire through visual analogue scale method
The level of the pain by questionnaire through visual analogue scale | day 7
  evaluation of the level of the pain by questionnaire through visual analogue scale method
Palliative 0-7 | immediately after surgery to 7 days later
  the number of palliatives the patient used during the first week after surgery
Pink aesthetic score | 3 months after surgery
  evaluation of the aesthetic score by photography
Pink aesthetic score | 6 months after surgery
  evaluation of the aesthetic score by photography

CONTACTS AND LOCATIONS:
Overall Officials: Neda Moslemi, Periodontist, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No